CLINICAL TRIAL: NCT04305535
Title: Clinical Trial to Evaluate the Effect of an Oligomeric Oral Nutritional Supplement on the Response in Intestinal Absorption and Inflammation, in Patients With CROHN Disease
Brief Title: Impact of an Oligomeric Diet in Intestinal Absorption and Inflammatory Markers in Patients With Crohn Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Adventia Pharma (Industry); Biopolis S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC032-19_FJD
Record Dates: First submitted 2020-03-05; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Crohn Disease; Absorption; Disorder, Protein; Absorption; Disorder; Absorption; Disorder, Fat; Absorption; Disorder, Carbohydrate; Malnutrition
Keywords: Oligomeric diet; Peptidic diet; Probiotics; Oral Nutritional Supplements
MeSH Terms: conditions — Crohn Disease; Platelet Glycoprotein IV Deficiency; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peptidic+Probiotic (Active Comparator): Nutritional intervention and dietary recommendations. Consumption of 2 tetra paks/day of a specific oral nutritional supplement and mix of probiotics during 6 months
  Interventions: Dietary Supplement: Peptidic+Probiotic
- Peptidic+Placebo (Active Comparator): Nutritional intervention and dietary recommendations. Consumption of 2 tetra paks/day of a specific oral nutritional supplement and placebo during 6 months
  Interventions: Dietary Supplement: Peptidic+Placebo
- Polymeric+Placebo (Placebo Comparator): Nutritional intervention and dietary recommendations. Consumption of 2 tetra paks/day of a specific oral nutritional supplement and placebo during 6 months
  Interventions: Dietary Supplement: Polymeric+Placebo

INTERVENTIONS:
Dietary Supplement: Peptidic+Probiotic — Oligomeric oral nutritional supplement (Bi1 peptidic) and a mix of probiotics
  * Bifidobacterium animalis subsp. lactis BPL1,
  * Lactobacillus rhamnosus BPL15,
  * Lactobacillus rhamnosus CNCM i-4036
  * Bifidobacterium longum ES1
  Arms: Peptidic+Probiotic
Dietary Supplement: Peptidic+Placebo — Oligomeric oral nutritional supplement (Bi1 peptidic) and a placebo
  Arms: Peptidic+Placebo
Dietary Supplement: Polymeric+Placebo — Polymeric oral nutritional supplement and a placebo
  Arms: Polymeric+Placebo

SUMMARY:
This is a randomized, multicenter, translational, triple-blind, clinical trial in patients with Crohn's disease, who will be prescribed an oral nutritional supplement to control symptoms in the acute phase and to recover in the remission phase.

DETAILED DESCRIPTION:
Multicentric, parallel, randomized, double blind and controlled clinical-nutritional study of 6 months of intervention and 3 study groups of treatment: Experimental group (peptidic diet with a mix of probiotics); Experimental group with placebo (peptidic diet with a placebo); and Control group (control with a polymeric nutritional oral supplement with a placebo) to evaluate the effect on the nutritional status, inflammatory markers and the intestinal absorption

ELIGIBILITY:
Inclusion Criteria:

* Unintentional weight loss of 5% in 6 months or a BMI less than 20kg/m2 or does not get the energy requirements with normal food.
* Willing to comply with the prescribed diet follow-up for CD.

Exclusion Criteria:

* Having received antibiotics in the previous 3 months
* Having undergone intestinal resection surgery≥70-75%
* Refuse to participate in the study
* Comorbidity that allows to suspect survival <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Malabsorption | 6 months
  Body Weight Change (kg)

SECONDARY OUTCOMES:
Changes in the consistency of the stools according to Bristol scale. | 6 months
  Bristol scale: type 1= separate hard lumps, type 2= sausage shaped but lumpy, type 3= like a sausage but with cracks on ots surface, type 4= like a sausage or sanake, smooth and soft, type 5= soft blobs with clear cut-edges, type 6= fluffy pieces with ragged edges, a mushy stool, type 7 = watery, no solid pieces.
Fat malabsorption | 6 months
  Presence of fat in the stool

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Aganzo-Yeves, RD, Principal Investigator — Hospital Universitario Fundación Jiménez Díaz; Clotilde Vázquez-Martínez, MD, Study Director — Hospital Universitario Fundación Jiménez Díaz
Locations (1):
- Miguel Aganzo Yeves, Madrid, Spain